CLINICAL TRIAL: NCT06907693
Title: The Effects of Drug Candidate CS1 on Lung Structure and Function Utilizing FRI, a Non-Invasive, Functional Respiratory Imaging System
Brief Title: The Effects of Drug Candidate CS1 on Lung Structure and Function Utilizing FRI
Status: Active, not recruiting | Type: Observational
Sponsor: Prisma Health-Upstate (Other)
Collaborators: Cereno Scientific AB (Industry)
Responsible Party: Sponsor
Other Study IDs: 2282898
Record Dates: First submitted 2025-03-27; First posted 2025-04-02 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: FLUIDDA FRI; FRI
MeSH Terms: conditions — Pulmonary Arterial Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CT Pulmonary Angiography Recipient: All subjects in this study will undergo CT pulmonary angiography scans at baseline (+/- 2 months from start of drug therapy), 4 months and 12 months.
  Interventions: Diagnostic Test: CT Pulmonary Angiography Scan

INTERVENTIONS:
Diagnostic Test: CT Pulmonary Angiography Scan — Computed tomography (CT) pulmonary angiography scan of the chest with IV contrast

SUMMARY:
Explore the impact of drug candidate CS1 on pathological vascular remodeling of small pulmonary arteries in the disease pulmonary arterial hypertension (PAH). This sub-study for CS1-004 aims to utilize FRI, an innovative, non-invasive imaging technology to visualize how long-term use of CS1 influences structural changes in pulmonary arteries. This sub-study seeks to provide valuable insights into the potential of CS1 to transform PAH treatment in some patients enrolled in the Expanded Access Program (CS1-004).

ELIGIBILITY:
Inclusion Criteria:

* Participation in the CS1-004 clinical trial

Exclusion Criteria:

* Inability to undergo a CT pulmonary angiography scan (i.e., claustrophobia)
* Individuals who are pregnant or who become pregnant during the sub-study
* eGFR <30 mL/min/1.73m2 as calculated by Modification of Diet in Renal Disease (MDRD)
* Allergy to Iodine contrast agents

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participation in the CS1-004 clinical trial at Prisma Health-Upstate
Sampling Method: Non-Probability Sample
Enrollment: 7 (Estimated)
Dates: Start 2025-03-14 (Actual); Primary Completion 2025-12-04 (Actual); Study Completion 2026-03-15 (Estimated)

PRIMARY OUTCOMES:
Ratio of BV5A to BV10A | From baseline CT scan to 12 month CT scan
  Change from baseline to month 12 in the ratio BV5A/BV10A

SECONDARY OUTCOMES:
Ratio of BV5A to BV5APR | From baseline CT scan to 12 month CT scan
  Change from baseline CT scan to 12 month CT scan regarding the ratio of the BV5A to BV5APR variable.
Ratio of BV5A to BV5APRA | From baseline CT scan to 12 month CT scan
  Change from baseline CT scan to 12 month CT scan regarding the ratio of the BV5A to BV5APRA variable.

CONTACTS AND LOCATIONS:
Locations (1):
- Prisma Health, Greenville, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] 1. US EPA O. Frequent Questions: Radiation in Medicine. www.epa.gov. Published December 4, 2023. https://www.epa.gov/radiation/frequent-questions-radiation-medicine